CLINICAL TRIAL: NCT04590066
Title: Testing Multiple Behavioral Science Strategies to Increase Flu-Shot Rates at a Large Retail Pharmacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 843523-Trial B
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Influenza, Human
Keywords: Influenza vaccination; behavioral science interventions; vaccination promotion
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the different arms.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: As treated participants will receive text messages, there is no scope for blinding. Care providers will not be made aware of subjects' participation in the study, or assigned treatment arms. The study team will only receive data on subjects' assigned arms and outcomes at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (23):
- Holdout control (No Intervention): Participants will only receive the standard pharmacy messaging.
- Unpacking Risks Treatment (Experimental): Participants will be asked to think about the risks of catching the flu this flu season and to respond with the location they are most likely to catch the flu out of a list of given options (e.g. at work, at home).
  Interventions: Behavioral: Flu shot text messages
- Unpacking Risks Control (Experimental): Participants will be asked to think about the risks of catching the flu this flu season and to respond to confirm that they have received the message.
  Interventions: Behavioral: Flu shot text messages
- Active Commitment Treatment (Experimental): Participants receive a gain framed notification that they are eligible for a flu shot. In addition, participants are told "Many people find it helpful to make a plan to get their shot" and are asked to commit by texting back "I will get a flu shot." Depending on their response, participants receive a general reminder or a commitment reminder 3 days later.
  Interventions: Behavioral: Flu shot text messages
- Active Commitment Control (Experimental): Participants receive a gain framed notification that they are eligible for a flu shot. Participants receive a general reminder 3 days later.
  Interventions: Behavioral: Flu shot text messages
- Self-Generated Social Norms Treatment (Experimental): Participants will first receive a message enjoining them to consider 2 peers who would want them to vaccinate. Then they will be asked to do those peers a favor by getting a vaccine at their next opportunity. They will receive a reminder 3 days later.
  Interventions: Behavioral: Flu shot text messages
- Self-Generated Social Norms Control (Experimental): articipants will be informed of the opportunity to receive a flu vaccine at their appointment. They will receive a reminder 3 days later.
  Interventions: Behavioral: Flu shot text messages
- Foot-in-the-Door Treatment (Experimental): Participants will first receive a message enjoining them to encourage someone else to receive a flu vaccine this year. They will then be given a message that they might copy-paste to forward to friends, thereby lowering the effort costs of messaging others. They will receive a reminder 3 days later.
  Interventions: Behavioral: Flu shot text messages
- Foot-in-the-Door Control (Experimental): Participants will be informed of the opportunity to receive a flu vaccine at their appointment. They will receive a reminder 3 days later.
  Interventions: Behavioral: Flu shot text messages
- Prosocial Condition (Experimental): Participants will receive a message describing the condition-specific benefit of getting a flu shot, and a reminder to ask for their flu shot. The message will also give prosocial reasons for vaccinating (i.e., protecting loved ones; preserving scarce resources).
  Interventions: Behavioral: Flu shot text messages
- Self-Oriented Condition (Experimental): Participants will receive a message describing the condition-specific benefit of getting a flu shot, and a reminder to ask for their flu shot.
  Interventions: Behavioral: Flu shot text messages
- Prosocial + COVID-19 (Experimental): Participants will receive a message describing the condition-specific benefit of getting a flu shot, and a reminder to ask for their flu shot. The message will also give prosocial reasons for vaccinating (e.g., protecting loved ones; preserving scarce resources). The message will also emphasize the pandemic (e.g., risk of hospital-acquired COVID-19 infection; wasting scarce resources).
  Interventions: Behavioral: Flu shot text messages
- Self-Oriented + COVID-19 (Experimental): Participants will receive a message describing the condition-specific benefit of getting a flu shot, and a reminder to ask for their flu shot. The message will also emphasize the pandemic (e.g., risk of hospital-acquired COVID-19 infection; wasting scarce resources).
  Interventions: Behavioral: Flu shot text messages
- Dynamic + Static Norm (Experimental): Participants will receive a text message encouraging them to get a flu shot and informing them that more American adults are getting their flu shot than ever before and how many Americans got their flu shot last year.
  Interventions: Behavioral: Flu shot text messages
- Dynamic Norm (Experimental): Participants will receive a text message encouraging them to get a flu shot and informing them that more American adults are getting their flu shot than ever before.
  Interventions: Behavioral: Flu shot text messages
- Dynamic Norms Control (Experimental): Participants will only receive a text message encouraging them to get a flu shot. They will not receive any norm information.
  Interventions: Behavioral: Flu shot text messages
- Sharing Humor (Experimental): Participants will receive a text message encouraging them to get the flu shot. The message will include a joke about the flu and will encourage participants to share the joke with nurses, doctors, or pharmacists.
  Interventions: Behavioral: Flu shot text messages
- Humor Placebo (Experimental): Participants will receive a text message encouraging them to get the flu shot. This message will include the same joke but participants will not be encouraged to share it.
  Interventions: Behavioral: Flu shot text messages
- No Humor Condition (Experimental): Participants will receive a text message encouraging them to get the flu shot.
  Interventions: Behavioral: Flu shot text messages
- Connecting the Past Self to the Future Self Treatment (Experimental): Participants will receive a text message prompt to recall the negative experience of getting sick. When asked, "Do you wish you could have avoided getting sick by getting a simple shot?", participants will have the chance to respond Y for yes or N for no. Regardless of their response, they will be prompted with a second text message to connect their past experience with present-day opportunities for preventative care (getting a flu shot) to protect the future self from the flu.
  Interventions: Behavioral: Flu shot text messages
- Connecting the Past Self to the Future Self Control (Experimental): In the first text message, participants will receive a simple text message encouragement to receive a flu shot. In the second text message, they will receive a reminder of the appointment time and provider name.
  Interventions: Behavioral: Flu shot text messages
- Reverse Inference Condition (Experimental): Participants will receive a text message encouraging them to get a flu shot and informing them that Americans who get flu shots are healthier, wealthier, and more educated.
  Interventions: Behavioral: Flu shot text messages
- Reverse Inference Control Condition (Experimental): Participants will receive a text message encouraging them to get a flu shot and informing them that Americans who get flu shots are less likely to get the flu.
  Interventions: Behavioral: Flu shot text messages

INTERVENTIONS:
Behavioral: Flu shot text messages — Participants will receive text messages per descriptions listed in the arms.
  Arms: Active Commitment Control; Active Commitment Treatment; Connecting the Past Self to the Future Self Control; Connecting the Past Self to the Future Self Treatment; Dynamic + Static Norm; Dynamic Norm; Dynamic Norms Control; Foot-in-the-Door Control; Foot-in-the-Door Treatment; Humor Placebo; No Humor Condition; Prosocial + COVID-19; Prosocial Condition; Reverse Inference Condition; Reverse Inference Control Condition; Self-Generated Social Norms Control; Self-Generated Social Norms Treatment; Self-Oriented + COVID-19; Self-Oriented Condition; Sharing Humor; Unpacking Risks Control; Unpacking Risks Treatment

SUMMARY:
This research aims to identify which behavioral science strategies are most effective at increasing flu vaccination rates overall and based on patients' individual characteristics. Past behavioral science interventions have shown promise in increasing flu vaccinations. For example, successful interventions have encouraged people to make concrete plans for when they will get a flu vaccination, sent automated calls or text messages reminding patients to get a flu vaccination , or provided financial incentives for getting vaccinated. Although these results are promising, these studies have been conducted in isolation on different populations, which makes it difficult to compare their interventions' effectiveness or to have enough power to reliably detect differing responses to interventions based on individual characteristics.

This research will simultaneously test 22 different SMS interventions to increase flu vaccinations compared to a holdout control condition in a "mega-study" and apply machine learning to identify which interventions work best for whom. The interventions are designed by behavioral science experts from the Behavior Change for Good Initiative (BCFG), Penn Medicine Nudge Unit (PMNU), and Geisinger Behavioral Insights Team (BIT). Customers of a large retail pharmacy who received a flu shot from the pharmacy last year and receive SMS notifications will be included in this study. We expect this to include approximately 1.2 million participants.

The specific aims of this research are to identify (1) which behavioral science strategies effectively increase flu vaccination rates overall, and (2) which strategies are most effective for different subgroups (e.g., based on age, gender, race).

ELIGIBILITY:
Inclusion Criteria:

1. Have agreed to receive SMS messages from the pharmacy
2. Received a flu shot from the pharmacy in the 2019-2020 flu season, as documented in their pharmacy records.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 734383 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Whether participants receive a flu shot vaccination at our pharmacy partner by December 31, 2020 | 98 days
  The primary outcome measure is whether participants receive a flu shot at our retail pharmacy partner by December 31, 2020 (as recorded in their pharmacy records) after receiving the SMS intervention on September 25, 2020.
  Participants who receive a flu shot before September 25, 2020 when they received the SMS intervention will be excluded from the analyses.

SECONDARY OUTCOMES:
Whether participants receive a flu shot vaccination at our pharmacy partner by October 31, 2020 | 37 days
  The secondary outcome measure is whether participants receive a flu shot at our retail pharmacy partner by October 31, 2020 (as recorded in their pharmacy records) after receiving the SMS intervention on September 25, 2020.
  Participants who receive a flu shot before they receive the SMS intervention on September 25, 2020 will be excluded from the analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutrona SL, Golden JG, Goff SL, Ogarek J, Barton B, Fisher L, Preusse P, Sundaresan D, Garber L, Mazor KM. Improving Rates of Outpatient Influenza Vaccination Through EHR Portal Messages and Interactive Automated Calls: A Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):659-667. doi: 10.1007/s11606-017-4266-9. Epub 2018 Jan 30. PMID 29383550
- [Background] Milkman KL, Beshears J, Choi JJ, Laibson D, Madrian BC. Using implementation intentions prompts to enhance influenza vaccination rates. Proc Natl Acad Sci U S A. 2011 Jun 28;108(26):10415-20. doi: 10.1073/pnas.1103170108. Epub 2011 Jun 13. PMID 21670283
- [Background] Regan AK, Bloomfield L, Peters I, Effler PV. Randomized Controlled Trial of Text Message Reminders for Increasing Influenza Vaccination. Ann Fam Med. 2017 Nov;15(6):507-514. doi: 10.1370/afm.2120. PMID 29133488
- [Background] Nowalk MP, Lin CJ, Toback SL, Rousculp MD, Eby C, Raymund M, Zimmerman RK. Improving influenza vaccination rates in the workplace: a randomized trial. Am J Prev Med. 2010 Mar;38(3):237-46. doi: 10.1016/j.amepre.2009.11.011. Epub 2009 Dec 24. PMID 20036102